CLINICAL TRIAL: NCT05352854
Title: In Vivo Morphological Changes of Ciliary Body and Trabecular Meshwork in High Myopia Eyes With Open-angle Glaucoma in Their Accommodation Induced by Pilocarpine
Brief Title: Morphological Changes of Ciliary Body and Trabecular Meshwork
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Myopia-OAG SSOCT
Record Dates: First submitted 2022-04-17; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma; Myopia
Keywords: ciliary body and trabecular meshwork
MeSH Terms: conditions — Glaucoma; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Health control (Experimental): emmetropia/low myopia (equivalent spherical lens > -3.00d, astigmatism ≤ 1.5d), best corrected visual acuity ≥1.0
  Interventions: Drug: 0.5% pilocarpine eye drops
- High myopia (Experimental): Equivalent spherical lens ≤-6.00D or axial length ≥26.5mm
  Interventions: Drug: 0.5% pilocarpine eye drops
- Primary open angle glaucoma (Experimental): emmetropia/low myopia (equivalent spherical lens > -3.00d, astigmatism ≤ 1.5d), diagnosed as POAG
  Interventions: Drug: 0.5% pilocarpine eye drops
- HM-POAG (Experimental): Equivalent spherical lens ≤-6.00D or axial length ≥26.5mm，diagnosed as POAG
  Interventions: Drug: 0.5% pilocarpine eye drops

INTERVENTIONS:
Drug: 0.5% pilocarpine eye drops — Subjects will be given 0.5% pilocarpine eye drops every five minutes for three times and wait for 40 minutes

SUMMARY:
Glaucoma is the leading cause of irreversible blindness worldwide. Although the pathogenesis remains unclear, pathologic increase in intraocular pressure (IOP) due to blocked aqueous outflow through the trabecular-Schlemm canal is known to be an important risk factor, and reduction of IOP is the only clinically validated way to retard the progression of OAG. Ciliary muscle plays a central role in the trabecular meshwork-Schlemm canal outflow pathway. Clinical evidence suggests that ciliary muscle contraction stimulated by cholinergic receptor agonist and retraction of ciliary body position after cataract surgery can dilate the lumen of Schlemm canal and reduce IOP. Currently, Ultrasound biomicroscopy (UBM) can obtain two-dimensional images of the anterior segment using high-frequency Ultrasound transducers in medical imaging studies of the ciliary body - trabecular meshwork -Schlemm canal complex. UBM has better tissue penetration than Optical coherence tomography (OCT) and can image the ciliary body better, but it has a lower resolution (30um to 50um) and is poor at imaging tiny tissues such as trabecular meshwork and Schlemm canal. The latest swept-source OCT (SS-OCT) has faster image capture rate (1000000 A scans/SEC), stronger penetration and higher resolution (8um axial resolution and 20um transverse resolution). The structure and morphology of ciliary body-trabecular meshwork-Schlemm canal complex can be clearly photographed. The investigators intend to use CASIA2 to image the ciliary body-trabecular meshwork-Schlemm canal complex before and after administration of pilocarpine in healthy individuals and patients with glaucoma to assess the effect of pilocarpine on the anatomy of the ciliary body-trabecular meshwork-Schlemm canal complex.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide. Although the pathogenesis remains unclear, pathologic increase in intraocular pressure (IOP) due to blocked aqueous outflow through the trabecular-Schlemm canal is known to be an important risk factor, and reduction of IOP is the only clinically validated way to retard the progression of OAG. Ciliary muscle plays a central role in the trabecular meshwork-Schlemm canal outflow pathway. When the ciliary muscle contraction, the elastic fiber network will pull trabecular meshwork away from Schlemm canal direction, trabecular meshwork and adjacent tissue gap increases, increasing aqueous outflow. Clinical evidence suggests that ciliary muscle contraction stimulated by cholinergic receptor agonist and retraction of ciliary body position after cataract surgery can dilate the lumen of Schlemm canal and reduce IOP. Currently, Ultrasound biomicroscopy (UBM) can obtain two-dimensional images of the anterior segment using high-frequency Ultrasound transducers in medical imaging studies of the ciliary body - trabecular meshwork -Schlemm canal complex. UBM has better tissue penetration than Optical coherence tomography (OCT) and can image the ciliary body better, but it has a lower resolution (30um to 50um) and is poor at imaging tiny tissues such as trabecular meshwork and Schlemm canal. The latest swept-source OCT (SS-OCT) has faster image capture rate (1000000 A scans/SEC), stronger penetration and higher resolution (8um axial resolution and 20um transverse resolution). The structure and morphology of ciliary body-trabecular meshwork-Schlemm canal complex can be clearly photographed. The novel anterior segment optical coherence tomography (AS-OCT) device, CASIA2 can accurately image the ciliary body-trabecular meshwork-Schlemm canal complex. The investigators intend to use CASIA2 to image the ciliary body-trabecular meshwork-Schlemm canal complex before and after administration of pilocarpine in healthy individuals and patients with glaucoma to assess the effect of pilocarpine on the anatomy of the ciliary body-trabecular meshwork-Schlemm canal complex.

ELIGIBILITY:
Inclusion Criteria:

* Emmetropia/low myopia,high myopia, primary open-angle glaucoma without high myopia, and high myopia with primary open-angle glaucoma
* have a good gaze to complete the test required inspection;

Exclusion Criteria:

* hypersensitivity to pilocarpine
* History of eye surgery, including cataract surgery, anti-glaucoma surgery, corneal surgery, retinal surgery, and eye trauma
* history of systemic diseases that may affect the eyes (such as diabetes, hypertension, etc.)
* intraocular chronic inflammatory diseases (uveitis, etc.), retinal diseases (retinal detachment, diabetic retinopathy, retinitis pigmentosa, etc.)
* Corneal scars and severe cataracts affect OCT imaging
* Eye diseases (angle-closure glaucoma, abnormal anterior segment development, neovascularization, etc.) that can affect trabecular meshwork and Schlemm canal structure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Morphology of ciliary body | baseline, pre-intervention(local application of pilocarpine eye drops)
  measurement of Morphology of ciliary body using CAISA2(The novel anterior segment optical coherence tomography (AS-OCT) device) and Image J software
Morphology of ciliary body | 40 minutes after the intervention(local application of pilocarpine eye drops)
  measurement of Morphology of ciliary body using CAISA2(The novel anterior segment optical coherence tomography (AS-OCT) device) and Image J software
Morphology of trabecular meshwork | baseline, pre-intervention(local application of pilocarpine eye drops)
  measurement of Morphology of trabecular meshwork using CAISA2(The novel anterior segment optical coherence tomography (AS-OCT) device) and Image J software
Morphology of trabecular meshwork | 40 minutes after the intervention(local application of pilocarpine eye drops)
  measurement of Morphology of trabecular meshwork using CAISA2(The novel anterior segment optical coherence tomography (AS-OCT) device) and Image J software

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Principal Investigator — Ophthalmology and Optometry Hospital